CLINICAL TRIAL: NCT06141798
Title: A Pragmatic Randomized Clinical Trial: Twice-weekly vs Thrice-weekly Incident hemoDialysis in Elderly Patients
Brief Title: Twice vs Thrice Weekly Incident Hemodialysis in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Soon Hyo Kwon, MD, Professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC21C0059
Record Dates: First submitted 2023-10-07; First posted 2023-11-21 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Age Problem; Dialysis; Complications; Frailty; Quality of Life
MeSH Terms: conditions — Frailty | interventions — Renal Dialysis

STUDY DESIGN:
Intervention Model Description: Pragmatic Randomization Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twice-weekly hemodialysis with incremental approach (Active Comparator)
  Interventions: Other: Hemodialysis
- Thrice-weekly hemodialysis (No Intervention)

INTERVENTIONS:
Other: Hemodialysis — Number of weekly hemodialysis treatment
  Arms: Twice-weekly hemodialysis with incremental approach

SUMMARY:
As Korea is becoming a super-aged society, the number of elderly patients with end-stage kidney disease (ESKD) is expected to increase rapidly. Therefore, the burden on Korean society will also increase.

Thrice-weekly hemodialysis is standard for renal replacement therapy. However, this regimen has not been validated for elderly ESKD patients with residual renal function. Elderly patients can have multiple comorbidities such as hypertension, diabetes, cardiovascular disease, and impaired physical activity. Frequent hemodialysis could provoke falls, hypotension, and cognitive impairment. Previous reports have suggested the potential benefit of twice-weekly hemodialysis with incremental increases in frequency when residual renal function decreases. In addition, twice-weekly hemodialysis decreases hospitalization rates in frail patients.

Therefore, the investigators hypothesized initiating renal replacement therapy with twice-weekly hemodialysis decreases the hopsitalizatoin rates compared with conventional thrice-weekly hemodialysis in elderly ESRD patients with residual renal function. This study is a pragmatic randomized clinical trial, multicenter study. Study subjects are incident ESRD patients (>= 60 years old, n=428) with residual urine volume ( > 500 mL/day) and follow up up to 2 years. Twice-weekly hemodialysis could be incremented according to clinical situations such as volume overload, hyperkalemia and uremic symptom. Primary outcome of this study is hospitalization rate during follow-up. Secondary outcomes include dialysis related hospitalization rate, the length of hospital stay, complication of dialysis,mortality rate and assessments of quality of life, frailty, and cost-utility.

DETAILED DESCRIPTION:
End-stage kidney disease (ESKD) poses a substantial public health challenge, with the number of patients requiring renal replacement therapy (RRT) globally reaching 2.61 million in 2010 and projected to rise to 5.43 million by 2030. In Korea, the incidence of hemodialysis (HD) has also been gradually increasing. The increase in HD incidence in South Korea is significantly linked to the aging population. Korea is one of the most rapidly aging countries in the world and the age of dialysis patients is also increasing, with more than half over the age of 60.

HD has potential advantages over conservative management or peritoneal dialysis in older adults, however, guidelines for optimal HD for the elderly have not yet been established. Typically, patients receive HD three times a week, with only a small proportion of patients receiving less frequent dialysis. However, potential disadvantages such as hemodynamic stress, vascular access problems, bleeding, falls and economic cost should be considered in older adults with ESKD.

In elderly patients, it is often difficult to maintain a thrice-weekly HD schedule due to the presence of other medical conditions and the challenges of frailty. Elderly patients have shown poor outcome even after initiation of HD. A study by Santos et al. demonstrated a more than twofold increased risk of mortality at 6 months in patients older than 75 years compared to those younger than 75. Another study using Japanese National Dialysis Registry data revealed a 30% mortality rate in those aged over 80 years within 1 year after initiation of HD, with frailty being one of the most important factors associated with early death after initiation of HD. Excessive HD in elderly patients can lead to malnutrition, low blood pressure during dialysis, poor quality of life, depression, and stress due to physical and temporal activity restriction. The increased risk of falls in HD patients is also a serious problem.

Incremental initiation of HD involves starting HD at a lower intensity than the standard 4 hours thrice weekly and gradually increasing the frequency and duration of dialysis as kidney function declines. The decision to initiate patients on incremental HD can be made based on clinical parameters such as urine volume or residual kidney function, socio-economic factors such as financial limitations or insurance coverage, or lack of availability of dialysis services. Current guidelines recommend that twice weekly dialysis be performed in patients with kidney urea clearance greater than 3ml/min/1.73m2 or a urine output over 0.5 liter per day.

A systemic review and meta-analysis showed no difference in mortality, hospitalization rates, or quality of life between patients receiving incremental and conventional HD, with improved preservation of residual renal function and a reduction in dialysis cost with incremental HD. One randomized controlled trial (RCT) showed no difference in episodes of fluid overload or hyperkalemia, but an increased risk of hyperkalemia with incremental HD. Another study showed lower hospitalization rate in incremental HD compared to conventional dialysis. These studies demonstrate the need for a large RCT comparing incremental and conventional HD.

However, current studies do not provide conclusive evidence on the benefits and risks of incremental HD in elderly patients. Therefore, the investigators are conducting a pragmatic RCT to determine whether the initiation of renal replacement therapy with twice-weekly HD reduces hospitalization rates compared to conventional thrice-weekly HD in older adults with ESKD.

Trial design PRIDE trial is designed as a pragmatic RCT comparing the effect of initiating twice-weekly hemodialysis with an incremental approach compared to thrice-weekly HD on hospitalization rates in elderly ESKD patients with RKF. A total of 428 participants will be recruited from 18 academic dialysis centers in Korea. Participants will have the flexibility to transfer to other dialysis centers as needed. The decision to increase dialysis frequency will be made by the treating physicians.

Hypothesis Our main hypothesis is that twice-weekly HD, when prescribed to older adults with RKF will reduce hospitalization rates compared with thrice-weekly HD.

1. Liyanage T, Ninomiya T, Jha V, et al. Worldwide access to treatment for end-stage kidney disease: a systematic review. Lancet 2015;385:1975-1982.
2. Hong YA, Ban TH, Kang CY, et al. Trends in epidemiologic characteristics of end-stage renal disease from 2019 Korean Renal Data System (KORDS). Kidney Res Clin Pract 2021;40:52-61.
3. Choi HS, Han KD, Oh TR, et al. Trends in the incidence and prevalence of end-stage renal disease with hemodialysis in entire Korean population: A nationwide population-based study. Medicine (Baltimore) 2021;100:e25293.
4. Verberne WR, Geers AB, Jellema WT, Vincent HH, van Delden JJ, Bos WJ. Comparative Survival among Older Adults with Advanced Kidney Disease Managed Conservatively Versus with Dialysis. Clin J Am Soc Nephrol 2016;11:633-640.
5. Corbett RW, Brown EA. Conventional dialysis in the elderly: How lenient should our guidelines be? Semin Dial 2018;31:607-611.
6. Bieber B, Qian J, Anand S, et al. Two-times weekly hemodialysis in China: frequency, associated patient and treatment characteristics and Quality of Life in the China Dialysis Outcomes and Practice Patterns study. Nephrol Dial Transplant 2014;29:1770-1777.
7. Santos J, Oliveira P, Malheiro J, et al. Predicting 6-Month Mortality in Incident Elderly Dialysis Patients: A Simple Prognostic Score. Kidney Blood Press Res 2020;45:38-50.
8. Yazawa M, Kido R, Ohira S, et al. Early Mortality Was Highly and Strongly Associated with Functional Status in Incident Japanese Hemodialysis Patients: A Cohort Study of the Large National Dialysis Registry. PLoS One 2016;11:e0156951.
9. Buemi M, Lacquaniti A, Bolignano D, et al. Dialysis and the elderly: an underestimated problem. Kidney Blood Press Res 2008;31:330-336.
10. Wang HH, Wu JL, Lee YC, et al. Risk of Serious Falls Between Hemodialysis and Peritoneal Dialysis Patients: A Nationwide Population-based Cohort Study. Sci Rep 2020;10:7799.
11. Caton E, Sharma S, Vilar E, Farrington K. Impact of incremental initiation of haemodialysis on mortality: a systematic review and meta-analysis. Nephrol Dial Transplant 2023;38:435-446.
12. Hemodialysis Adequacy Work G. Clinical practice guidelines for hemodialysis adequacy, update 2006. Am J Kidney Dis 2006;48 Suppl 1:S2-90.
13. Kalantar-Zadeh K, Unruh M, Zager PG, et al. Twice-weekly and incremental hemodialysis treatment for initiation of kidney replacement therapy. Am J Kidney Dis 2014;64:181-186.
14. Vilar E, Kaja Kamal RM, Fotheringham J, et al. A multicenter feasibility randomized controlled trial to assess the impact of incremental versus conventional initiation of hemodialysis on residual kidney function. Kidney Int 2022;101:615-625.
15. Murea M, Patel A, Highland BR, et al. Twice-Weekly Hemodialysis With Adjuvant Pharmacotherapy and Transition to Thrice-Weekly Hemodialysis: A Pilot Study. Am J Kidney Dis 2022;80:227-240 e221.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Clinical diagnosis of end stage kidney disease
* Starting maintenance hemodialysis within one month
* 24-hour urine output ≥ 500 ml at randomization
* Sufficient understanding of the study procedures and requirements.

Exclusion Criteria:

* Left ventricular ejection fraction < 40%)
* Liver cirrhosis
* Current treatment for an active malignancy or active infection
* Onability or refusal to provide written informed consent
* enrollment in another clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | Follow up: 2 years
  The total number of hospitalizations per 100 person-years

SECONDARY OUTCOMES:
Dialysis related hospitalization rate | Follow up: 2 years
  The total number of dialysis hospitalizations per 100 person-years
Length of Hospital Stay | Follow up: 2 years
  per 1000 person-days
Complication of dialysis | Follow up: 2 years
  Any complication of dialysis associated
Mortality rate | Follow up: 2 years
  Any cause of death
The Clinical Frailty Scale | Follow up: 2 years
  One item, minimum point: 1, maximum point: 9, High scores means worse outcome
Cost effective | Follow up: 2 years
  Incremental Cost-Effectiveness Ratio, Higher scores means better
Kidney Disease Quality of Life Instrument (KDQOL) | Follow up: 2 years
  24 items, minimum point 1, maximum point 5, high score means worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Soon Hyo Kwon, MD, Principal Investigator — Soonchunhyang University Hospital
Locations (7):
- South Korea (7):
  - Soonchunhyang University Hospital Bucheon, Bucheon-si
  - Hallym University Medical Center- Chuncheon, Chuncheon
  - Soonchunhyang University Seoul Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Koera University Guro Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han M, Jeon H, Yu BC, Song SH, Chung S, Lim C, Sohn H, Noh JW, Kwon SH. A Pragmatic Randomized clinical trial: twice-weekly vs. thrice-weekly Incident hemoDialysis in Elderly patients (PRIDE): study protocol. Kidney Res Clin Pract. 2026 Jan;45(1):130-139. doi: 10.23876/j.krcp.23.177. Epub 2023 Dec 18. PMID 38148125